CLINICAL TRIAL: NCT02939378
Title: Ketogenic Diet Adjunctive to Salvage Chemotherapy for Recurrent Glioblastoma:a Pilot Study
Acronym: KGDinrGBM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Song Lin (Other)
Responsible Party: Sponsor-Investigator, Song Lin, Proffessor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0009
Record Dates: First submitted 2016-10-06; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Glioblastoma Multiforme
Keywords: ketogenic diet; recurrent glioblastoma; chemotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketogenic diet group (Experimental): Ketogenic diet adjuvant to salvage chemotherapy was given to recurrent glioblastoma. Blood glucose and ketone were kept more than 2mmol/L during salvage chemotherapy. The side effect was observed and recorded. Tumor volume was monitored and the efficacy was recorded.
  Interventions: Dietary Supplement: Ketogenic diet
- Standard diet group (Other): Standard diet adjuvant to salvage chemotherapy was given to recurrent glioblastoma. Blood glucose and ketone were recorded during salvage chemotherapy. The side effect was observed and recorded. Tumor volume was monitored and the efficacy was recorded.
  Interventions: Dietary Supplement: Standard diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet adjuvant to salvage chemotherapy is given to recurrent glioblastomas.
  Arms: ketogenic diet group
Dietary Supplement: Standard diet — Standard diet adjuvant to salvage chemotherapy is given to recurrent glioblastomas.
  Arms: Standard diet group

SUMMARY:
Recently, ketogenic diet has been recognized a useful treatment strategy for glioblastoma in vitro.

Therefore, the purpose of the study is to evaluate the safety and efficacy of ketogenic adjuvant to salvage chemotherapy for recurrent glioblastoma.

DETAILED DESCRIPTION:
Diet change by limiting carbohydrates and increasing the proportion of fatty acids and proteins can lead to ketogenic metabolism and might limit energy production in tumor cells and inhibit tumor growth.

In a pilot of recurrent glioblastoma, ketogenic diet adjuvant salvage chemotherapy was given as interventional group and standard diet adjuvant salvage chemotherapy was given as control group.

The study examines whether a ketogenic diet adjunctive to salvage chemotherapy can be applied to the patients and may inhibit tumor growth and influence the quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. Karnovsky Performance Score of 60 or more.
3. histologically confirmed glioblastoma multiforme, grade 4
4. Ability and willingness to signed informed consent form.
5. Documented recurrence or progression after surgical resection/debulking, radiation and temozolomide chemotherapy.
6. normal function of liver and kidney

Exclusion Criteria:

1. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, carnitine deficiency and pancreatitis
2. History of uncontrolled hyperlipidemia or hyperglycemia.
3. History of human immunodeficiency virus, or hepatitis C
4. Pregnancy or breastfeeding
5. Inability or unwillingness of subject to give written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Effects | one year
  Number of participants with treatment-emergent adverse effects while on ketogenic diet.

SECONDARY OUTCOMES:
The Chemosensitivity of Tumor | one year
  MRI(Magnetic Resonance Imaging) will be used to measure changes in brain tumor size (cm^2).
Overall Survival | one year
  Participants were followed until reported death
Ketosis | one year
  Urine and blood ketosis (mmol/L) were measured
Quality of Life | one year
  quality of life measured by the Karnofsky Performance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Song Lin, M.D.,, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided